CLINICAL TRIAL: NCT04569097
Title: Defining Novel Pharyngeal Pressure Metrics to Predict Dysphagia Treatment Outcomes and Clinical Prognosis Using High-resolution Manometry
Brief Title: Novel Pharyngeal Metrics to Predict Dysphagia Outcomes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: N3221-R
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Dysphagia; Swallowing Disorders
Keywords: dysphagia; manometry; swallowing; veterans
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Patients will be stratified into the following groups: Group A) Patient Group receiving Pharyngeal strengthening (n=150); and Group B) Healthy Controls (n=50). Participants' age may range from 18-99 years old, however, the investigators expect most study participants will be >60 years old due to the age range typically affected by dysphagia.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient group (Experimental): lingual strengthening
  Interventions: Other: standard of care lingual strengthening
- Controls (No Intervention): No history of dysphagia (swallowing disorder) or minimal to mild dysphagia not requiring a strengthening program

INTERVENTIONS:
Other: standard of care lingual strengthening — standard or care lingual strengthening approaches with outcome measured with novel pressure metrics
  Arms: Patient group

SUMMARY:
This multi-site trial will follow a cohort of Veterans with dysphagia for 8 weeks as they undergo clinically guided oropharyngeal exercises with oropharyngeal strengthening as the primary goal. Veterans with dysphagia will be assessed at three time points: baseline, 4 weeks after treatment initiation, and 8 weeks after treatment initiation. A non-dysphagic Veteran control group will also undergo data collection at parallel time points, without completion of a treatment paradigm. The investigators will then compare patients to non-dysphagic controls using manometry, videofluoroscopy, diet assessment, functional reserve tests, and patient-reported outcome measures.

The investigators aim to 1) quantify change in pressure measures of swallowing function resulting from dysphagia treatment; 2) determine which combination of standard of care and/or pressure-based metrics best track with outcome measures; and 3) develop multimodal prognostic algorithms that predict treatment success. This research will establish a precise outcome measurement paradigm suitable for dysphagia clinical care and research, thus improving clinical confidence and paving the way for a personalized medicine approach for dysphagia rehabilitation in Veterans.

DETAILED DESCRIPTION:
This multi-center trial will follow a cohort of Veterans with dysphagia for 8 weeks as they undergo clinically guided oropharyngeal exercises with oropharyngeal strengthening as the primary goal. Veterans with dysphagia will be assessed at three time points: baseline, 6-4 weeks post-treatment, and 8 weeks post-treatment. A non-dysphagic Veteran control group (n=50) will also undergo data collection at parallel time points, without completion of a treatment paradigm. The investigators will then compare patients to nondysphagic controls using pHRM, videofluoroscopy, diet assessment, functional reserve tests, and patient reported outcome measures. The investigators aim to 1) quantify change in pHRM measures of swallowing function resulting from dysphagia treatment; 2) determine which combination of standard of care and/or pHRM-based metrics best track with patient-reported outcome measures; and 3) develop multimodal prognostic algorithms that predict treatment success. This research will establish a precise outcome measurement paradigm suitable for dysphagia clinical care and research, thus improving clinical confidence and paving the way for a personalized medicine approach for dysphagia rehabilitation in Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Signed an informed consent form
* Receive a dysphagia diagnosis by a speech-language pathologist
* Must have a dysphagia treatment plan with the goal of strengthening the oropharyngeal musculature
* English speaking

Exclusion Criteria:

* history of allergic response to barium
* history of allergic response to topical anesthetics

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
pHRM pressure change | Baseline, 4 weeks, and 8 weeks
  Will assess the change in pressure by pharyngeal high resolution manometry over the time frame The primary measure of interest is Integral Pressure during the 10 mL swallow at the tongue base Range is From: 0 mmHg*sec, no pressure recorded to up to 250 mmHg*sec., very high pressures recorded, normal range is age and sex dependent Range (114+/-50 to167 +/-80) Positive change would be a movement toward normal range of pressure. This metric is measured automatically in both Software systems used to evaluate pharyngeal pressure (WiscMano and Swallow gateway)
Swallowing clinical and fluoroscopic change | Baseline, 4 weeks, and 8 weeks
  Will assess the change in fluoroscopy and clinical assessments over the time frame The primary tool of measurement is the combined score of the MBSImP this is a 17 item standardized tool to measure impairment of swallow identified using contrast barium swallows. We will use the composite pharyngeal score which ranges from 0 to 3, the higher the score the more abnormal the swallow function, Normal swallows will score 5 or less and severe dysphagia will score 9 or higher.
  Movement toward 0 is a positive or improved swallow function, movement toward 23 is negative or worsening swallow function
Patient reported outcome changes | Baseline, 4 weeks, and 8 weeks
  Sydney swallowing questionnaire (SSQ) The SSQ is a patient reported symptom scale with 17 questions, each scaled from 0+ no dysfunction to 100 equal extreme dysfunction using a 100mm visual analogue scale with 0 and 100 as anchors. the total score can be recorded for 0 to 1700, Normal swallowers will average 40 with a range of 200 to 0, Dysphagia patients average 800 with a range of 150 to 1600. Movement toward 0 will be considered an improvement, movement toward 1700 worsening in swallowing ability preserved by the patient.

SECONDARY OUTCOMES:
Patient reported outcome changes | Baseline, 4 weeks, and 8 weeks
  Eating assessment tool -10, The Eat 10 is a short 10 question swallowing assessment tool 10 questions each scaled 0 to 4, total can be between 0 and 40.
  The normal swallowers will score under 2. The mean (+/- SD) EAT-10 score of the normal cohort was 0.40 +/- 1.01.
  The mean EAT-10 score for those with oropharyngeal dysphagia, 23.10 +/- 12.22 Changes toward 0 will be identified as improved swallow symptom function, changes toward 40 worsening symptoms
Patient reported outcome changes, Diet change | Baseline, 4 weeks, and 8 weeks
  International Dysphagia Diet Standardization initiative, Functional Oral intact scale Standardize scale of diet (liquid and solid food) iddsi.org foods scaled from regular diet 7 to liquidized 3, and liquids scaled from thin liquids 0 to extremely think 4 Improvement in diet will be report if patients move toward 0 in liquid intake and toward 7 in solid food intact and movement in the opposite directions will be evidence of poorly food and liquid tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M. McCulloch, MD, Principal Investigator — William S. Middleton Memorial Veterans Hospital, Madison, WI
Locations (3):
- United States (3):
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/97/NCT04569097/ICF_000.pdf